CLINICAL TRIAL: NCT00486928
Title: Twenty-five-year Experience With the Medtronic-Hall Valve Prosthesis
Acronym: Hall-Kaster
Status: Completed | Type: Observational
Sponsor: Oslo University Hospital (Other)
Other Study IDs: 06/8009
Record Dates: First submitted 2007-06-14; First posted 2007-06-15 (Estimated); Last update posted 2011-07-25 (Estimated); Status verified 2011-07

CONDITIONS: Aortic Valve Disease
Keywords: Valves, heart disease, prosthesis.
MeSH Terms: conditions — Aortic Valve Disease; Heart Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- AVR: All consecutive patients in the study period

SUMMARY:
Background-:. The Medtronic-Hall (MH) valve was developed and for the first time implanted in Oslo in 1977. A total of 1,104 patients received this valve at Rikshospitalet-Radiumhospitalet HF in the period 1977-87. In the present study we followed all 816 patients undergoing aortic valve replacement (AVR) over a 25-year period.

DETAILED DESCRIPTION:
The Medtronic-Hall (MH) tilting valve disk was first implanted in Oslo in June 1977. From 1977 through 1987, the valve was used as the only valve of choice and inserted in a total of 1,104 consecutive patients at our department.

The MH valve is made of a single piece of titanium with no welds. The disk is made of tungsten impregnated graphite with a carbon pyrolytic coating. The tungsten renders the disk radiopaque. In the aortic position the maximal opening is 75˚. A central aperture in the disk allows free rotation. The valve is rotatable in the sewing ring. The sewing ring is made of Teflon. Aortic sizes are 20-31 mm (outer diameter).

The initial clinical results were published in 1979 (1). The cohort of patients has been followed-up and analysed at 5, 10 and 15 years (2-5). In the present study we report our 25-year follow-up data for the 816 patients undergoing aortic valve replacement (AVR) with special reference to survival, functional status, valve-related complications and the impact of concomitant surgery.

ELIGIBILITY:
Inclusion Criteria:

* All patients with aortic valve replacement 1977-87

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All consecutive patients undegoing AVR during inclusion period
Sampling Method: Probability Sample
Enrollment: 816 (Actual)
Dates: Start 2004-05; Study Completion 2005-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jan L Svennevig, MD,PhD, Principal Investigator — Rikshospitalet, Oslo
Locations (1):
- Rikshospitalet, Oslo, Norway